CLINICAL TRIAL: NCT02544425
Title: Phase II Study of VIDL (VP-16, Ifosfamide, Dexamethasone, L-asparaginase) Chemotherapy Followed by High-dose Chemotherapy and Autologous Stem Cell Transplantation in Patients With Stage III/IV Extranodal NK-T-Cell Lymphoma
Brief Title: VP-16, Ifosfamide, Dexamethasone, L-asparaginase Chemotherapy in Patients With Extranodal Natural Killer T Cell Lymphoma (VIDL+ASCT)
Acronym: VIDL+ASCT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Seog Kim, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-05-035
Record Dates: First submitted 2015-09-06; First posted 2015-09-09 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Extranodal NK-T-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — Etoposide; Ifosfamide; Dexamethasone; Asparaginase; Busulfan; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VIDL+ASCT (Experimental): 1. VIDL Induction (repeated 28 days) : VP-16, Ifosfamide, Dexamethasone, L-asparaginase
  2. Peripheral blood stem cell mobilization:Etoposide
  3. Conditioning regimen for autologous stem cell transplantation:Busulfan,Melphalan,Etoposide
  Interventions: Drug: Etoposide; Drug: Ifosfamide; Drug: Dexamethasone; Drug: L-asparaginase; Drug: Busulfan; Drug: Melphalan

INTERVENTIONS:
Drug: Etoposide — Subjects will receive Etoposide 100 mg/m2 + 5% dextrose in water 500 mL intravenous over 90 mins D1-3 of VIDL chemotherapy. After that, Etoposide will be administered 375mg/m2 D1-2 with G-colony stimulating factor (10 ug/kg) injection in step of Peripheral Blood Stem Cell Collection. Also It will be administered 400mg/m2 on conditioning regimen.
  Other Names: VP-16
Drug: Ifosfamide — It will be administered1.2g/m2 + 5% dextrose in water 100 mL intravenous over 1 hr D1-3
Drug: Dexamethasone — It will be administered 40mg/day PO or IV D1-3
Drug: L-asparaginase — It will be administered 4000 IU/m2 intramuscular D8, 10, 12, 14, 16, 18, 20
Drug: Busulfan — Conditioning regimen for autologous stem cell transplantation:
  Busulfan 3.2 mg/kg D -8, -7, -6
Drug: Melphalan — Conditioning regimen for autologous stem cell transplantation:
  Melphalan 70 mg/m2 D -3, -2

SUMMARY:
Open-labeled, multicenter phase II study of VIDL (VP-16, Ifosfamide, Dexamethasone, L-asparaginase) chemotherapy followed by high-dose chemotherapy and autologous stem cell transplantation in patients with stage III/IV extranodal NK/T-cell Lymphoma.

DETAILED DESCRIPTION:
Extranodal NK/T cell lymphoma (ENKTL) is a rare and aggressive lymphoma subtype, but standard front-line therapy has not been established. The clinical outcome of patients (pts) with ENKTL after the treatment of conventional chemotherapy, especially pts with advanced stage, was generally poor. Therefore, high-dose chemotherapy followed by autologous stem cell transplantation (ASCT) as a consolidation could be one of promising strategies to improve the outcome of ENKTL. However, there have been few studies reporting the survival outcome or prognostic significances of front-line ASCT in pts with ENKTL. Thus, the aim of this study was to investigate the outcome of patients with advanced-stage ENKTL who had undergone front-line ASCT.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed extranodal NK/T cell lymphoma
* Aged between 19 and 65 years
* Previously untreated history
* Performance status: Eastern Cooperative Oncology Group 0-2
* Ann Arbor stage III and IV
* At least one in positron emission tomograph(PET)/CT positive lesion or in 2-dimensional computerized tomography

  * mass lesions more than 2 cm by conventional CT or more than 1 cm by spiral CT
  * Skin lesions or physically detected mass more than 2 cm
* Cardiac ejection fraction ≥ 45 % as measured by multiple gated acquisition scan(MUGA) or 2D echogram(ECHO) without clinically significant abnormalities
* Adequate liver functions: Transaminase (AST/ALT) < 3 X upper normal value(or < 5 x upper limit of normal in the presence of NK/T lymphoma involvement of the liver)
* Bilirubin < 2 X upper normal value(or < 5 x upper limit of normal in the presence of DLBCL involvement of the liver)
* Serum Creatinine < 2.0 mg/dL
* Adequate bone marrow functions: hemoglobin ≥ 9 g/dL absolute neutrophil count (ANC) ≥ 1,500/μL and platelet count ≥ 75,000/μL, unless abnormalities are due to bone marrow involvement by lymphoma
* Expected life is more than 180 days (more than 6 months)
* A negative serum or urine pregnancy test prior to treatment must be available both for pre-menopausal women and for women who are < 1years after the onset of menopause. Premenopausal women should be treated with appropriate contraception such as hormone contraception, intra-uterine device, spermicidal condom and etc. during and one month after the treatment.
* Voluntarily signed the informed consent including fully understand of clinical procedures and processing steps for the clinical trial

Exclusion Criteria:

* Patients who have serious medical condition, abnormal laboratory results or psychiatric problems
* Other subtypes non-Hodgkin's lymphoma than NK/T cell lymphoma
* Patients who have aggressive NK/T cell leukemia
* NK/T cell lymphoma with Primary Central Nervous System (CNS) involvement. However, patients who have only had prophylactic intrathecal chemotherapy against CNS disease are eligible.
* Patients with a known history of HIV seropositivity or hepatitis C virus (HCV) (+). Patients who have carrier hepatitis B virus (HBV) (+) are eligible. However, primary prophylaxis using antiviral agents is recommended for HBV carrier to prevent HBV reactivation during whole treatment period.
* Any other malignancies within the past 5 years except curatively treated non-melanoma skin cancer or in situ carcinoma of cervix uteri
* Pregnant or lactating women, women of childbearing potential not employing adequate contraception
* Other serious illness or medical conditions i. Unstable cardiac disease despite treatment, myocardial infarction within 6 months prior to study entry ii. History of significant neurologic or psychiatric disorders including dementia or seizures iii. Active uncontrolled infection (viral, bacterial or fungal infection) iv. Other serious medical illnesses
* Concomitant administration of any other experimental drug under investigation, or concomitant chemotherapy, hormonal therapy, or immunotherapy.
* Serious allergy history for experimental drugs
* Patients who contraindication to the study drug use

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2016-02-21 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | 2 years

SECONDARY OUTCOMES:
objective overall response rate | 2 years
Number of subjects with Adverse Events as a Measure of safety and tolerability | 2 years
overall survival | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: won-Seog Kim, MD,Ph.D, Principal Investigator — Samsung Medical Center
Locations (2):
- South Korea (2):
  - Samsung Medical Center, Seoul, Seoul, Korea, Republic of
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Yes